CLINICAL TRIAL: NCT05435534
Title: Effect of a Multicomponent Intervention With Telerehabilitation and Vivifrail on Functional Capacity After Hip Fracture: a Randomized Control Trial
Brief Title: Effect of a Multicomponent Intervention on Functional Capacity After Hip Fracture
Acronym: ActiveFLS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacion Miguel Servet (Other)
Collaborators: Hospital of Navarra (Other); NavarraBiomed Biomedical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ActiveFLS
Record Dates: First submitted 2022-05-25; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Hip Fractures; Osteoporosis; Fall; Frailty Syndrome; Rehabilitation
MeSH Terms: conditions — Hip Fractures; Osteoporosis; Frailty

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multicomponent intervention (Experimental): Participants randomly assigned to the Multicomponent intervention group will received a multifactorial intervention.
  Interventions: Other: ActiveFLS intervention
- Usual care group (Active Comparator): Participants randomly assigned to the usual care group will received normal outpatient care, including physical rehabilitation when needed.
  Interventions: Other: Usual care group

INTERVENTIONS:
Other: ActiveFLS intervention — * A comprehensive geriatric assessment with a multicomponent physical exercise program guideline based on ActiveHip+ for 3 months. In the subsequent revisions, exercise guidelines from the Vivifrail program will be given
  * A protocolized nutritional intervention will be carried out. In case of oral nutritional supplementation, supplements enriched in β-hydroxy-β-methylbutyrate (HMB) will be selected
  * Osteoporosis treatments according to national guideline
  * A review and adaptation of the treatment will be carried out according to the STOPP (Screening Tool of Older Persons' Prescriptions) and START (Screening Tool to Alert to Right Treatment) criteria
  * An approach will be made to the patient's mood and fear of falling. In case of depression, both pharmacological and non-pharmacological approaches will be assessed
  * Screening for cognitive impairment will be performed. In the event of evidence of memory problems, a recommendations for cognitive stimulation will be delivered
  Arms: Multicomponent intervention
Other: Usual care group — Participants randomly assigned to the usual care group will receive normal outpatient care, including physical rehabilitation when needed.
  Arms: Usual care group

SUMMARY:
Due to the clinical, functional, cognitive and social complexity of older adults after fragility hip fractures (defined as those produced by low-impact trauma), the investigators propose an intervention.

This intervention involves a multidisciplinary and multicomponent program consisting of physical exercise with tele-rehabilitation, nutritional assessment and other variables related to comprehensive geriatric assessment.

The investigators want to improve functional status, quality of life and prevent new fractures. In addition, the investigators try to optimize treatments and resources based on the functional status of patients and their life expectancies, improving care and healthcare cost

DETAILED DESCRIPTION:
Study aims

1. Improve functional capacity (Short Physical Performance Battery, SPPB) in older patients with fragility hip fractures through a multidisciplinary and multicomponent program and increase the quality of life (EuroQol-5 Dimension) and reduce the use of resources (admission and readmission to emergency department or in-hospital) at 3, 6 and 12 months compare with usual care
2. Analyze the subgroups of patients that benefit the most from the respective interventions, identifying factors of the patient (sociodemographic, clinical, functional and cognitive) and of the intervention (type of exercise, nutritional supplementation, pain control, etc.), which could explain differences in the effectiveness of the intervention at 3, 6 and 12 months
3. Analyze the effect of multidisciplinary and multicomponent intervention in older adults with hip fracture on cognitive capacity (4-AT, MMSE), risk of falls (number of falls, Falls Efficacy Scale), depression (GDS), pain (VAS), polypharmacy, geriatric syndromes and nutritional status (MNA) compare with usual care at 3, 6 and 12 months
4. Developmentally monitor the changes achieved through the intervention, as well as the factors that determine the perpetuation of the benefits of the long-term.
5. Examine the effect of a multi-component program on muscle mass (DXA), bone formation and resorption (BTMs) at 12 months
6. Estimate the prevalence of frailty, multimorbidity and geriatric syndromes in older adults with fragility hip fracture and the changing at 3, 6 and 12 months.
7. Estimate the use of resources necessary to carry out the intervention program, as well as the average time to carry out the comprehensive geriatric assessment, and which is the most cost/efficient tool in this case.
8. Examine the applicability of a tele-rehabilitation program (ActiveHip) in older adults with hip fracture.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 75 years.
* Diagnosis of frailty hip fracture (those produced by low-impact trauma).
* Absence of terminal-stage disease
* Barthel scale score ≥ 60 points.
* Previous independence for wandering measured as FAC ≥6
* Capability/Support for using ActiveHip+ app

Exclusion Criteria:

* Moderate-severe cognitive impairment considered as a Goldberg Global Deterioration Scale score ≥ 5.
* Refusal to sign the informed consent by the patient / main caregiver / legal guardian or inability to obtain it
* Secondary osteoporosis
* Nursing home

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2022-05-26 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB) | T1 Baseline T2 1month T3 3 months T4 6 months T5 12 months
  The primary endpoint will be the changes measured at baseline and follow-up

SECONDARY OUTCOMES:
Barthel index | T1 Baseline T2 1month T3 3 months T4 6 months T5 12 months
  Barthel Index of independence during activities of daily living (ADLs). This index ranges from 0 worst to 100 best The endpoint will be the changes measured at baseline and follow-up
FAC scale | T1 Baseline T2 1month T3 3 months T4 6 months T5 12 months
  The Functional Ambulation Categories (FAC) is a functional walking test that evaluates ambulation ability. This index ranges from 0 worst to 5 best
  The endpoint will be the changes measured at baseline and follow-up
GDS scale | T1 Baseline T2 1month T3 3 months T4 6 months T5 12 months
  Global Deterioration Scale of Reisberg (GDS Reisberg). GDS Reisberg describes 7 clinically distinguishable global stages, from normality (GDS 1) to severe dementia (GDS 7) of the Alzheimer disease.
  The endpoint will be the changes measured at baseline and follow-up
Number of Participants with Institutionalization | T2 1month T3 3 months T4 6 months T5 12 months
  The endpoint will be the new Number of Participants with institutionalization
  The endpoint will be the changes measured at follow-up
Hand grip stength | T1 Baseline T2 1month T3 3 months T4 6 months T5 12 months
  Hand grip strength was measured following the Gronigen Elderly Test using a Smedley Hand Dynamometer. The best of three attempts (with 30 seconds rest between each attempt) was recorded.
  The endpoint will be the changes measured at baseline and follow-up
Rate of Frailty | T1 Baseline T2 1month T3 3 months T4 6 months T5 12 months
  Fried frailty index . This scores range from 0-5 (i.e., 1 point for each component; 0=best to 5=worst) and represent frail (3-5), pre-frail (1-2), and robust (0)
  The endpoint will be the changes measured at baseline and follow-up
Lawton index | T1 Baseline T2 1month T3 3 months T4 6 months T5 12 months
  Lawton index of independence durante instrumental activities of daily living. This index ranges from 0 worst to 8 best
  The endpoint will be the changes measured at baseline and follow-up
Mini- Mental State Examination (MMSE) | T1 Baseline T2 1month T3 3 months T4 6 months T5 12 months
  MMSE is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. This index ranges from 0 worst to 30 best The endpoint will be the changes measured at baseline and follow-up
Changes in the quality of life measured by the Spanish version of the EuroQol-5 Dimension (EQ-5D) questionnaire | T1 Baseline T2 1month T3 3 months T4 6 months T5 12 months
  The endpoint will be the changes measured at baseline and follow-up
  The EQ records the respondent's overall current health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine' Minimum 0 Maximum 100 Higher scores mean a better outcome
Mini Nutritional Assessment (MNA) | T1 Baseline T2 1month T3 3 months T4 6 months T5 12 months
  Scale to diagnosis of malnutrition. This index ranges from 0 worst to 30 best
  The endpoint will be the changes measured at baseline and follow-up
Mortality | T2 1month T3 3 months T4 6 months T5 12 months
  The endpoint will be incidence of this event
Admission and readmission to hospital | T2 1month T3 3 months T4 6 months T5 12 months
  The endpoint will be incidence of this event
New fractures | T2 1month T3 3 months T4 6 months T5 12 months
  The endpoint will be incidence of this event

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Martinez-Velilla, PhD, Study Director — Fundación Instituto de Investigación Sanitaria de Navarra
Locations (1):
- Hospital Universitario de Navarra (HUN), Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: Yes
We plan to share data under reasonable request
Supporting Information: Study Protocol